CLINICAL TRIAL: NCT06308679
Title: A Bioequivalence Study of Two Formulations of 10-mg Empagliflozin Tablets in Healthy Thai Volunteers Under Fasting Conditions
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pharma Nueva (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: BE 001-24
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Healthy Vollunteer
Keywords: Empagliflozin; Bioequivalence study
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Generic Empagliflozin 10 mg tablets (Experimental): Generic Empagliflozin 10 mg tablets (test drug)
  Interventions: Drug: Empagliflozin 10 mg tablets; Drug: JARDIANCE®
- ARDIANCE® (Active Comparator): ARDIANCE® (Empagliflozin 10 mg tablets (reference drug))
  Interventions: Drug: Empagliflozin 10 mg tablets; Drug: JARDIANCE®

INTERVENTIONS:
Drug: Empagliflozin 10 mg tablets — Empagliflozin 10 mg tablets (test drug)
Drug: JARDIANCE® — Empagliflozin 10 mg tablets (reference drug)
  Other Names: Empagliflozin 10 mg tablets

SUMMARY:
Objectives:

Primary:

to evaluate the bioequivalence of two formulations of Empagliflozin tablets, test formulation and reference innovator formulation, after a single oral dose administration in healthy Thai subjects under fasting conditions

Secondary:

To examine the pharmacokinetics and safety of test and reference formulations

Study Design:

A Bioequivalence Study of Two Formulations of 10-mg Empagliflozin Tablets in Healthy Thai Volunteers under Fasting Conditions

DETAILED DESCRIPTION:
Subjects will be fasted at least 10 hours before dosing. After that a single dose of 10-mg Empagliflozin tablets will be administered along with 240 mL of drinking water under fasting condition. In each period, a total of 21 blood samples (approximately 6 mL each) from 21 sampling time points will be collected at pre-dose (6-mL tubes) and at 0.33, 0.67, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 14.00, 24.00, 36.00 and 48.00 h post dose. Blood glucose level will be measured at approximately pre-dose, 0.33, 0.67, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00 hours post-dose in each period for subject's safety. During blood sample collection, one drop of blood will be used for this test.

ELIGIBILITY:
Inclusion Criteria:

1. Thai male and/or female age between 18-55 years
2. Has body mass index (BMI) between 18.0-30.0 kg/m2
3. Has been determined healthy by physical examination, assessment of medical history, and vital signs (blood pressure (systolic blood pressure not lower than 90 or not over 139 mmHg, diastolic blood pressure not lower than 60 or not over 89 mmHg), body temperature, pulse rate, respiratory rate) or showing no clinically significant abnormalities in the opinion of principal investigator or designated physicians
4. Has normal or acceptable results (being assessed as not clinically significant by the clinical investigator) for all screening tests including: Complete Blood Count (CBC), Fasting Blood Sugar (FBS), Aspartate Aminotransferase (AST or SGOT), Alanine Aminotransferase (ALT or SGPT), Alkaline Phosphatase (ALP), Total Bilirubin, Blood Urea Nitrogen (BUN), Creatinine (Cr), Potassium, Sodium, Chloride, Phosphate and Urinalysis
5. Has negative result for Hepatitis B viral profile (HBsAg)
6. Has normal or acceptable report (being assessed as not clinically significant by the clinical investigator) for EKG
7. Male subjects agree to use effective contraceptive from screening visit to the follow-up visit.
8. Female subjects must agree not to become pregnant for the entire participation period and must have a negative result for a urine pregnancy test performing at screening and prior to dosing at period 1 and period 2.
9. Female subjects who is childbearing potential and using effective non-hormonal contraceptive methods (e.g., condom, diaphragm, cervical cap or sexual abstinence) or total abstinence from sexual intercourse from screening visit to the follow-up visit.
10. Female subject who is non-childbearing potential (hysterectomy, both ovaries removed, surgically sterilized or postmenopausal (for at least 12 consecutive months of amenorrhea)).
11. Non-smokers (never smoked or no smoking within the previous 1 year)
12. Refrain from using herbal medications, cannabis containing products, dietary supplements (e.g., St. John's Wort, ginkgo biloba, garlic supplements), vitamins, grapefruit or grapefruit juice, or pomelo within 14 days before the first administration of study drug (Day 1). Subjects must agree to refrain from these items until the last collection time-point of period 2.
13. Subjects must have ended the systematic medications at least 30 days prior to Day 1 and agree to continue their refraining throughout the follow-up period.
14. Subjects must refrain from drinking caffeine and alcohol for at least 72 hours prior to Day 1 and agree to continue their refraining throughout the last collection time-point of period 2.
15. Has ability and intention to comply with the requirement of study and available for the whole study period
16. Willing to participate and voluntarily signed the informed consent form prior to participate the study

Exclusion Criteria:

1. Known hypersensitivity to empagliflozin and/or related structure and/or its constituents.
2. Has history or concurrent symptoms of cardiovascular, gastrointestinal, hematological disorders, renal and hepatic impairment and/or any disease that may affect the bioavailability of the drug.
3. Alcohol abuse or excessive use (more than 1 time/week) in the last 12 months
4. Alcohol breath test at screening visit or before admission show alcohol concentration more than 0.000 %BAC.
5. History of drug abuse or urine sample shows a positive test for Morphine, Tetrahydrocannabinol and Methamphetamine at screening visit or before admission.
6. Following a special diet (e.g., vegetarian) or dieting one month before the study initiation.
7. A pregnant woman (positive pregnancy test at screening or prior to dosing in each period) or woman in breast feeding period
8. A woman of childbearing potential and using hormonal contraceptive methods including oral contraceptives, hormone replacement therapy and transdermal contraceptives within 14 days prior to dosing and during the entire period of the study and/or using injected, intrauterine and implanted hormonal methods of contraception within 3 months prior to dosing and during the entire period of the study
9. A participant in any investigation drug study within last 30 days prior to screening (from the last visit that received medication to the screening visit)
10. Has blood donated within last 2 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-05-28 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-07 (Estimated)

PRIMARY OUTCOMES:
Plasma area Under the Curve (AUC(0-48hr)) for Empagliflozin | Through 48 hours post dose
  Plasma area Under the Curve (AUC(0-48hr)) for Empagliflozin
Peak Plasma Concentration (Cmax) of Empagliflozin | 48 hours post dose
  Peak Plasma Concentration (Cmax) of Empagliflozin

CONTACTS AND LOCATIONS:
Overall Officials: Porranee Puranajoti, Principal Investigator — International Bio service

IPD SHARING:
Plan to Share IPD: No
Confidential